CLINICAL TRIAL: NCT02615990
Title: Impact of the Erigo Machine on Functional Recovery in ICU
Brief Title: Impact of the Erigo Machine on Functional Recovery in ICU Patients
Acronym: Mobility
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Vendor equipment agreement expired
Sponsor: Lisa J. Fryman (Other)
Responsible Party: Sponsor-Investigator, Lisa J. Fryman, Nursing Director Trauma/Surgical Services, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Erigo 15-0519
Record Dates: First submitted 2015-11-05; First posted 2015-11-26 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Trauma Patients Requiring Physical Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Erigo Pro plus standard Physical Therapy (Experimental): The Erigo device therapy is a combination of tilt table with robotic stepper device allowing for cyclic leg loading. It also includes Functional Electrical Stimulation to optimize active neuromuscular stimulation. It will be used once a day to replace one of the standard PT therapies. The exercise mimics walking beyond what regular range of motion provides. Patients will have 2 additional PT therapies 20 minutes of standard range of motion movements.
  Interventions: Device: Erigo Pro
- Standard Physical Therapy (Active Comparator): Patients will have 3 standard Physcial Therapy session. Patients will have 2 additional PT therapies 20 minutes of standard range of motion movements.
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Device: Erigo Pro — Verticalization table with two integrated robotic devices for leg movement and cyclic loading
  Other Names: Verticalization table; Item #29673 Hocoma products
  Arms: Erigo Pro plus standard Physical Therapy
Other: Standard Physical Therapy — Patients receive standard physical therapy.
  Arms: Standard Physical Therapy

SUMMARY:
This study will assess the effects of the Erigo applied as part of the early mobilization program in the Trauma ICU at the University of Kentucky. It is our hypothesis, that with the Erigo, critically ill patients will tolerate verticalization and mobilization earlier and safely resulting in improved outcomes measured by increased mobility and strength on ICU discharge, decreased requirements for mechanical ventilation, reduced complication rates and decreased ICU and hospital LOS.

DETAILED DESCRIPTION:
The "Erigo" by Hocoma is a combination of tilt table with a robotic stepper device allowing for cyclic leg loading. Erigo now also includes Functional Electrical Stimulation to optimize active neuromuscular stimulation. It allows for protected gradual verticalization and mobilization based on patient tolerance and progress. It has been shown to improve orthostatic tolerance, cerebral blood flow and muscle strength.

Prospective Randomized Controlled Trial will compare two groups. The patients that meet inclusion criteria will be randomized into either the treatment group or a control group. General ICU mobility guidelines consist of scaled activity related to the patients' stability. The control group will get the general ICU mobility treatments and the treatment group will have one mobility treatment replaced with the Erigo treatment.

ELIGIBILITY:
Inclusion Criteria: Admission to Trauma ICU

1. Trauma Patients requiring physical therapy (including severe traumatic brain injury or polytrauma without extremity fractures or unstable thoracic or lumbar spine fracture
2. Burn patients requiring physical therapy
3. GI surgery patients requiring physical therapy
4. Necrotizing fasciitis patient requiring physical therapy

Exclusion Criteria:

Patients with the following conditions:

1. Non-weight bearing on lower extremities
2. Untreated DVT
3. Active hemorrhage
4. Leg length >102cm or <72cm
5. Weight >135kg
6. Systolic BP > 20mmHg sustained for 10min
7. Heart rate >20bpm outside goal for more than 20min
8. Intracranial pressure (ICP) >20mmHg sustained for 10min if applicable,
9. Temperature >38.2C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bernard, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
This study did not gather data beyond one intervention before closing. This is not applicable.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — study terminated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Tolerance During Verticalization
Description: Rapid decreases in blood pressure are a common clinical challenge when trauma patients go from lying down to standing. Changes in blood pressure will be compared between groups to determine if verticalization with an ERIGO Pro tilt table will alleviate the drop in blood pressure more quickly than standard of care. Participants will have their blood pressure measured upon initial verticalization after injury and at each treatment session there after until they achieve ambulation (the ability to move without assistance). Data will be presented as the number of days of treatment required to achieve blood pressure homeostasis during the positional change from lying to standing.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Orthostatic Tolerance During Ambulation
Description: Rapid decreases in blood pressure are a common clinical challenge when trauma patients go from standing to full ambulation. Changes in blood pressure will be compared between groups to determine if verticalization with an ERIGO Pro tilt table will alleviate the drop in blood pressure more quickly than standard of care. Participants will have their blood pressure measured upon initial unassisted standing and then during each treatment session there after until discharge. Data will be presented as the number of days of treatment required to achieve blood pressure homeostasis during the positional change from standing to full ambulation.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: ICU Length of Stay
Description: The duration of stay in the Trauma ICU will be measured and compared between groups. Data will be presented as mean number of days in the ICU.
Time Frame: Up to three months
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Description: The duration of hospitalization will be measured and compared between groups. Data will be presented as mean number of days the participant is hospitalized.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Pneumonia While Hospitalized
Description: Incidence of pneumonia while hospitalized will be determined by clinical symptoms to include temperature >100.8 degrees F, WBC>12,000 WBC/mm3 , PaO2/Fio2 ratio < 300 mmHg, positive respiratory culture for organisms and chest x-ray indicative of pneumonia. Total incidence will be compared between groups and presented as a total count of pneumonia diagnoses per group.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Urinary Tract Infections While Hospitalized
Description: Incidence of urinary tract infection during hospitalization will be determined by clinical symptoms to include temperature of > 100.8 degrees F, WBC> 12000 WBC/MM3, patient complaints of pain, positive urine culture. Total incidence will be compared between groups and presented as a total count of urinary tract infection diagnoses per group.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Deep Vein Thrombosis (DVT)
Description: Incidence of DVT with be determined based on clinical symptoms to include pain and positive duplex ultrasound or other diagnostic tool
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Incidence of Pressure Ulcers
Description: Incidence of pressure ulcers determined by physical observation. Total incidence will be compared between groups and presented as a total count of pressure ulcer diagnoses per group.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Incidence of Physical Instability
Description: Incidence of physical instability with be calculated as the number of falls per participant while hospitalized. Data will be presented as the number of falls per participant per group.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Catheter Disruption
Description: Incidence of unplanned removal/displacement of lines/tubes/catheters. Data will be presented as the number of disruptions per participant per group.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Measure of Physical Capacity
Description: Kansas University Hospital Physical Therapy Acute Care Functional Outcome Tool will be utilized to assess the participant's overall physical function prior to discharge. . Total score: 0 - 32, usually divided by 25%, 50%, >75% (minimum, moderate, maximum functionality). The higher the score, the great physical function the participant has.
Time Frame: At discharge (up to 1 year)
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Measure of Muscle Power
Description: The Muscle Research Council Muscle Scale will be used to determine actual muscle power generation vs the anticipated power generation prior to discharge. Total score: 0 - 5, 5 is normal muscle function. Data are presented as units on a scale.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Fall Risk
Description: Participant fall risk will be determined prior to discharge using the Berg Balance Scale to assess impairment of balance function through the completion of several functional tasks. The data are presented as units on a scale. The higher the number the lower the fall risk.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Assessment of Participant Mobility
Description: The ICU Mobility Scale ranks a participant's mobility on a scale of 0-32, were a score of zero is a completely non-mobile individual and a score of 32 is a fully ambulatory individual. Data will be collected at the time of discharge. The data are presented as units on a scale.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Independent Ambulation
Description: The number of hospital days required for the participant to regain independent ambulation (the ability to walk 5 meters unassisted) with be measured and presented as total days.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Mid-leg Muscle Circumference
Description: Mid-leg muscle circumference will be measure using a metric tape measure at hospital admission and again just prior to discharge. Data will be presented as the change in muscle circumference (cm) over time.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Patients Discharged From Hospital to Home
Description: The number of participants discharged to their home will be counted and presented as a percentage of the total participants in that arm.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Patients Discharged From Hospital to Skilled Nursing Facility
Description: The number of participants discharged to a skilled nursing home will be counted and presented as a percentage of the total participants in that arm.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Patients Discharged From Hospital to a Long Term Care Facility
Description: The number of participants discharged to a long term care facility will be counted and presented as a percentage of the total participants in that arm.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Patients Discharged From Hospital to an Acute Rehabilitation Facility
Description: The number of participants discharged to am acute rehabilitation facility will be counted and presented as a percentage of the total participants in that arm.
Time Frame: Up to one year
Population: ERIGO Pro manufacture requested the device be returned before any subject completed the protocol
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during hospitalization, up to one year.
Arm/Group | Erigo Pro Plus Standard Physical Therapy | Standard Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated by the device manufacturer prior to any subject completing the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No